CLINICAL TRIAL: NCT07350499
Title: Long-Term CLinical Evaluation of Aspiration ThRombectomy Using the Symphony or ProdIgy Thrombectomy System - CLEAR-IT
Brief Title: Aspiration Thrombectomy Using the Symphony or Prodigy System
Acronym: CLEAR-IT
Status: Recruiting | Type: Observational
Sponsor: Imperative Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ICI-2025-002
Record Dates: First submitted 2025-11-21; First posted 2026-01-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Arterial Thromboembolism; Venous Thromboembolism; Pulmonary Embolism
Keywords: Pulmonary Embolism; Thrombus; Thromboembolism; Aspiration; Aspiration thrombectomy; Anticoagulation; Peripheral vasculature
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism; Thrombosis; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Peripheral Arterial: Subjects in this cohort will undergo aspiration thrombectomy to remove thrombus from the peripheral arterial vasculature
  Interventions: Device: Prodigy Thrombectomy System
- Peripheral Venous: Subjects in this cohort will undergo aspiration thrombectomy to remove thrombus from the peripheral venous vasculature
  Interventions: Device: Symphony Thrombectomy System
- Pulmonary Embolism: Subjects in this cohort will undergo aspiration thrombectomy to remove thrombus from the pulmonary vasculature
  Interventions: Device: Symphony Thrombectomy System

INTERVENTIONS:
Device: Prodigy Thrombectomy System — Removal of thrombus/emboli from blood vessels in the peripheral vasculature
  Groups: Peripheral Arterial
Device: Symphony Thrombectomy System — Removal of thrombus/emboli from blood vessels in the peripheral vasculature
  Groups: Peripheral Venous
Device: Symphony Thrombectomy System — Removal of thrombus/emboli from the pulmonary vasculature
  Groups: Pulmonary Embolism

SUMMARY:
The study is designed to evaluate the short-term and long-term clinical performance and safety of the Symphony and Prodigy thrombectomy systems used in endovascular procedures across the peripheral or pulmonary vasculature.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age
2. Subject is willing and able to comply with the follow-up schedule specified in this protocol
3. Subject is willing and able to provide written informed consent prior to any study-related data collection
4. Subject has a planned procedure, involving the use of Imperative Care vascular devices within their intended use

Exclusion Criteria:

1. Subjects with any contraindications per the applicable Instructions for Use
2. Subject with life expectancy of less than 1 year
3. In the opinion of the Investigator, the patient is not a suitable candidate for intervention with Imperative Care devices
4. Subject who may be unable to complete study follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll subjects aged 18 years and older who are undergoing endovascular procedures in the peripheral or pulmonary vasculature systems where, in the opinion of the treating physician, Imperative Care devices are appropriate for use within their cleared indications. All subjects must meet the general eligibility criteria and provide written informed consent prior to any study-specific data collection.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2026-01-23 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Peripheral Arterial Cohort | 30 days
  Freedom from major (above-ankle) unanticipated amputation of the index limb
Peripheral Venous Cohort | 30 days
  Target venous patency defined as patent flow in the treated segment without ≥50% restenosis or re-occlusion, no reintervention and no re-thrombosis as assessed by duplex ultrasound or venography
Pulmonary Embolism (PE) Cohort | 30 Days
  Mean change in the tricuspid annular plane systolic excursion to pulmonary artery systolic pressure ratio (TAPSE/PASP) from baseline, measured on transthoracic echocardiography (TTE) and independently adjudicated

SECONDARY OUTCOMES:
Peripheral Arterial Cohort | 90 Days
  Freedom from major (above-ankle) amputation of the index limb
Peripheral Arterial Cohort | 180 Days
  Freedom from major (above-ankle) amputation of the index limb
Peripheral Arterial Cohort | 30 Days
  Major adverse cardiovascular events (MACE) rate
Peripheral Arterial Cohort | 90 Days
  Major adverse cardiovascular events (MACE) rate
Peripheral Arterial Cohort | 180 Days
  Major adverse cardiovascular events (MACE) rate
Peripheral Arterial Cohort | 30 Days
  Target vessel patency assessed using change in ankle-brachial index
Peripheral Arterial Cohort | 90 Days
  Target vessel patency assessed using change in ankle-brachial index
Peripheral Arterial Cohort | 180 Days
  Target vessel patency assessed using change in ankle-brachial index
Peripheral Arterial Cohort | 30 Days
  Target vessel patency assessed using change in Rutherford claudication grade
Peripheral Arterial Cohort | 90 Days
  Target vessel patency assessed using change in Rutherford claudication grade
Peripheral Arterial Cohort | 180 Days
  Target vessel patency assessed using change in Rutherford claudication grade
Peripheral Arterial Cohort | 30 Days
  Rate of re-intervention for index limb due to re-thrombosis
Peripheral Arterial Cohort | 90 Days
  Rate of re-intervention for index limb due to re-thrombosis
Peripheral Arterial Cohort | 180 Days
  Rate of re-intervention for index limb due to re-thrombosis
Peripheral Arterial Cohort | 90 Days
  Quality of life assessment using Vascular Quality of Life Questionnaire-6 (VascuQOL-6)
Peripheral Arterial Cohort | 180 Days
  Quality of life assessment using Vascular Quality of Life Questionnaire-6 (VascuQOL-6)
Peripheral Arterial Cohort | 30 Days
  All-cause mortality
Peripheral Arterial Cohort | 90 Days
  All-cause mortality
Peripheral Arterial Cohort | 180 Days
  All-cause mortality
Peripheral Venous Cohort | Intraprocedural
  Technical success defined as complete or near complete (>75%) reduction in Marder score from baseline to immediately after the use of the device and prior to any use of adjunctive device, as independently adjudicated
Peripheral Venous Cohort | 48 hours
  Rate of Major Adverse Events (MAEs) as adjudicated by an independent medical monitor and defined as the occurrence of any of the following:
  * Major bleeding
  * Device-related mortality
  * Device-related Serious Adverse Events (SAE)
Peripheral Venous Cohort | Hospital Discharge
  Re-thrombosis of the treated venous segment, confirmed by imaging in accordance with institutional standards of care, associated with recurrent symptoms or requiring reintervention after the index procedure and before hospital discharge
Peripheral Venous Cohort | 90 Days
  Proportion of patients demonstrating decrease in Villalta score
Peripheral Venous Cohort | 180 Days
  Proportion of patients demonstrating decrease in Villalta score
Peripheral Venous Cohort | 180 Days
  Target venous patency, defined as patent flow in the treated segment without ≥50% restenosis or re-occlusion, no reintervention and no re-thrombosis as assessed by duplex ultrasound or venography
Peripheral Venous Cohort | 180 Days
  Quality of life and symptom severity assessment using the Venous Insufficiency Epidemiological and Economic Study (VEINES -QOL)
Peripheral Venous Cohort | 30 Days
  All-cause mortality
Peripheral Venous Cohort | 90 Days
  All-cause mortality
Peripheral Venous Cohort | 180 Days
  All-cause mortality
Pulmonary Embolism Cohort | Intraprocedural
  Change in pulmonary artery pressure
Pulmonary Embolism Cohort | 48 hours
  Mean change in tricuspid annular plane systolic excursion (TAPSE) / pulmonary artery systolic pressure (PASP) ratio from baseline, measured on transthoracic echocardiography (TTE) and independently adjudicated
Pulmonary Embolism Cohort | 48 hours
  Rate of Major Adverse Events (MAEs) as adjudicated by an independent medical monitor and defined as the occurrence of any of the following:
  * Major bleeding
  * Device-related mortality
  * Device-related Serious Adverse Events (SAE)
Pulmonary Embolism Cohort | 48 hours
  Right ventricle to left ventricle (RV/LV) ratio reduction from baseline
Pulmonary Embolism Cohort | 30 days
  Right ventricle to left ventricle (RV/LV) ratio reduction from baseline
Pulmonary Embolism Cohort | 90 Days
  Proportion of patients with improved or unchanged New York Hearth Association (NYHA) functional class
Pulmonary Embolism Cohort | 180 Days
  Proportion of patients with improved or unchanged New York Hearth Association (NYHA) functional class
Pulmonary Embolism Cohort | 30 Days
  Pulmonary Embolism recurrence
Pulmonary Embolism Cohort | 90 Days
  Pulmonary Embolism recurrence
Pulmonary Embolism Cohort | 180 Days
  Pulmonary Embolism recurrence
Pulmonary Embolism Cohort | 30 Days
  Quality of life assessed by the Pulmonary Embolism Quality of Life (PEmb-QoL) questionnaire
Pulmonary Embolism Cohort | 90 Days
  Quality of life assessed by the Pulmonary Embolism Quality of Life (PEmb-QoL) questionnaire
Pulmonary Embolism Cohort | 180 Days
  Quality of life assessed by the Pulmonary Embolism Quality of Life (PEmb-QoL) questionnaire
Pulmonary Embolism Cohort | 30 Days
  All-cause mortality
Pulmonary Embolism Cohort | 90 Days
  All-cause mortality
Pulmonary Embolism Cohort | 180 Days
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Steven Abramowitz, MD, Principal Investigator — Medstar Health Research Institute; Maya Serhal, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Huntsville Hospital, Huntsville, Alabama, United States

IPD SHARING:
Plan to Share IPD: No